CLINICAL TRIAL: NCT05123183
Title: The Effect of Acupressure and Back Massage on Lactation in Cesarean Deliveries: A Randomized Controlled Trial
Brief Title: Nonpharmacological Methods and Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, resmiye kaya odabaş, research assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Resmiye-01
Record Dates: First submitted 2021-10-23; First posted 2021-11-17 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Lactation
Keywords: lactation; cesarean delivery; acupressure; back massage
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Active Comparator): Acupressure will be applied to ST36 and CV17 points.
  Interventions: Other: acupressure group
- Back Massage (Active Comparator): Back massage will be applied.
  Interventions: Other: back massage group
- Control Group (Active Comparator): No application will be made to the mothers in this group, and the amount of milk will be measured by weighing the baby before and after breastfeeding.
  Interventions: Other: control group

INTERVENTIONS:
Other: acupressure group — A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position of the mother, leaving the application points exposed. The most preferred points ST36 and CV17 were selected from the points reported to affect lactation by reviewing the literature on the points to be compressed. Acupressure will be applied to CV17 point (single point) and ST36 point (bidirectional, right and left) for 2 minutes for a total of 6 minutes. Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it will be moved to the other point in the symmetrical region and the application will be made without interruption. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch.
  Arms: Acupressure group
Other: back massage group — The mother sits in the chair and leans forward, placing her arms on the table at her level and resting her head on her arms. The mother's breasts are naked and freely released. The researcher massages the mother from top to bottom on both sides of the spine between the scapula bones. At this time, his fists are clenched and the thumb is open. While pressing firmly with his fists, small circular friction movements are made with his thumb. From the neck to the scapula, both sides of the spine are rubbed at the same time for 3 minutes. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch.
  Arms: Back Massage
Other: control group — No application will be made to the mothers in this group, and the amount of milk will be measured by weighing the baby before and after breastfeeding.
  Arms: Control Group

SUMMARY:
Primiparous mothers after cesarean section often encounter insufficient milk production during breastfeeding. This study was planned as a randomized controlled study to examine the effect of acupressure and back massage on lactation in cesarean deliveries. The research will be carried out between July 2021 and July 2023 with mothers who had a cesarean section at Kocaeli University Research and Application Hospital and Health Sciences University Derince Training and Research Hospital. The research will be carried out with three groups as acupressure, back massage and control group. The sample number was calculated using the G*Power 3.1.9.2 program and the acupressure group: 24, the back massage group: 24, and the control group: 24. In order to increase the analysis power, the number of samples was increased by 25% and n=30 for each group (acupressure group: 30, back massage group: 30, and control group: 30). It is planned to collect the data with the Introductory Information Form, the Newborn Follow-up Form, the Mother's Follow-up Form, and the Visual Analogue Scale by which the Mothers Evaluate Lactation Onset Symptoms. The mothers will be given acupressure 4 minutes acupressure group, back massage group 3 minutes back massage, and no application will be made to the control group, once in the post-op 0th day, 2 times in the post-op 1st day and once in the post-op 2nd day. 15 minutes after the applications, the baby will be weighed while hungry and will be breastfed under the control of the researcher. Babies will be weighed again after breastfeeding. The data of the research will be evaluated using the Statistical Package for the Social Sciences 20.0 program. In the evaluation of the data; descriptive statistics will be given as percentage, arithmetic mean±standard deviation, median and minimum-maximum values, independent two-sample t-test for normally distributed variables and Mann-Whitney U test for non-normally distributed variables. Repeated measure covariance analysis will be applied to reveal the difference between the milk amounts of the mothers between the groups. Statistical significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Objective: The aim of this study is to examine the effects of acupressure and back massage on lactation in cesarean deliveries.

Hypotheses:

H01: There is no difference in the amount of breast milk between the acupressure, back massage group and the control group in cesarean deliveries.

H02: There is no difference between the acupressure, back massage group and the control group in terms of lactation onset symptoms in cesarean deliveries.

This study was designed as a randomized controlled experimental study. The study was carried out in Kocaeli University Research and Application Hospital and Health Sciences University Derince Training and Research Hospital obstetrics service between July 2021 and July 2023. planned to be carried out.

Primiparous mothers who performed cesarean section at Kocaeli University Research and Application Hospital and Health Sciences University Derince Training and Research Hospital will constitute the research population. The sample size was calculated based on the research conducted by Arumsari et al. 2018 to examine the effect of acupressure and relaxation exercise combination on breast milk production and breastfeeding self-efficacy. The sample size of the study was calculated using the G*Power 3.1.9.2 program and the mean, standard deviation and sample size values of the breast milk variable included in the related article were taken into account in calculating the effect size. The mean and standard deviation values of the breast milk variable in the experimental group were 30.1±16.9 and n=12. In the control group, the mean and standard deviation values of the breast milk variable were 17.6±7.4 and n=12. The effect size was calculated as 0.47 by using the mean, standard deviation and sample number values of the related article. The minimum number of individuals to be included in the sample of this study was calculated by taking G*Power 3.1.9.2 and effect size: 0.47, α= 0.05, power: 0.95, and the sample size was at least 72 mothers (n= 24 for each group). ) was determined. In order to increase the analysis power, the number of samples was increased by 25% and n=30 for each group (acupressure group: 30, back massage group: 30, and control group: 30). The random number generation program in which group the mothers included in the study would be in was determined from the website called "Research Team Generator" and divided into three groups. Thus, each mother's group number was determined and recorded. Thus, each mother's number and group number would be determined and recorded.

Data Collection Tools Introductory Information Form: This form was prepared by the researcher in line with the literature. The form includes 38 questions including socio-demographic, obstetric characteristics, information about general health, and characteristics related to breast milk and breastfeeding.

Newborn Follow-up Form: It contains introductory information about the newborn, weight follow-up, feeding frequency and number of stools, and bilirubin values. Within the scope of the study, blood will not be taken from the newborn, and the existing bilirubin values will be used.

Mother Follow-up Form: This form, prepared by the researcher, contains the estimated amount of milk according to the difference in weight of the baby in the morning and evening, the average daily sleep duration of the mother and the amount of fluid consumed by the mother.

The Visual Analog Scale by which the Mothers Evaluate Lactation Onset Symptoms: The Visual Analog Scale used in the study of Mauri et al. 2015 will be used in the assessment. Tension, temperature increase and pain in the breasts, which are the signs of starting lactation, will be scored between 0-10. 0 "None", 1-2 "Too little", 3-4 "A little too much", 5-6 "Too much", 7-8 "Too much" and 9-10 "Too much, unbearable" and what is the total score? it will be understood that the higher the lactation initiation symptoms, the more.

Pre-Application In order to assess whether the questions have been understood, a preliminary study will be conducted with five mothers before starting the study. As a result of the evaluation, it will be evaluated whether there is a need for editing in the data forms and adjustments will be made. Those included in the preliminary study will not be included in the sample group.

Data Collection After obtaining the permissions of the ethics committee and the institution, the study can be performed by going to the institutions and performing a cesarean section between the first 8-12 hours on the 0th postoperative day. Mothers who are between working hours will be welcomed. Mothers who meet the research criteria will be informed about the purpose, content and method of the research and those who want to participate in the research will be determined.

To mothers;

* 1 time on post-op day 0,
* Post-op 1st day 2 times,
* Acupressure and back massage will be applied 4 times in total, once on the 2nd post-op day. No application will be made to the control group.

If the baby weighing process;

* Post-op 2 times on day 0,
* Post-op 1st day 4 times,
* Post-op will be done 2 times on the 2nd day, 8 times in total. After 15 minutes (min) of the applications, the baby will be weighed and breastfed while hungry (before breastfeeding). It will be weighed again to measure the average value of the amount of breast milk taken immediately after breastfeeding. The scale will have a sensitivity of 5 grams and will be provided by the researcher.

Acupressure Application Technique A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position for the mother, leaving the application points exposed. The most preferred points ST36 and CV17 were selected from the points reported to affect lactation by examining the literature on the points to be applied. Acupressure will be applied to CV17 point (single point) and ST36 point (bidirectional, right and left) for 2 minutes for a total of 6 minutes. Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it will be moved to the other point in the symmetrical region and the application will be made without interruption. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch.

The assistant researcher received acupressure training on 13.05.2021 and the principal researcher also has acupressure training.

Acupressure Application Points:

ST 36 point: The Stomach Meridian 36 point is located on the front of the leg and above the tibialis anterior muscle. It increases blood flow and plays a role in milk production.

CV17: Conception Vessel 17 point is located between the nipples, in the midline of the sternum, in the 4th intercostal space. This point stimulates blood circulation and stimulates milk production.

Back Massage Application Technique:

The mother sits in the chair and, leaning forward, puts her arms on the table at her level and rests her head on her arms. The mother's breasts are naked and freely released. The researcher massages the mother from top to bottom on both sides of the spine between the scapula bones. At this time, his fists are clenched and the thumb is open. While pressing firmly with his fists, small circular friction movements are made with his thumb. From the neck to the scapula, both sides of the spine are rubbed at the same time for 3 minutes. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch.

Evaluation of Data The data of the study will be evaluated using the Statistical Package for the Social Sciences (SPSS) 22.0 program. All data will first be evaluated with Kolmogorov-Smirnov for conformity to normal distribution and then analyzed according to fitness for normal distribution. For descriptive statistics, percentages will be used in general, arithmetic mean±standard deviation for those that are suitable for normal distribution, median and minimum-maximum values for those that are unsuitable. Comparisons between groups for numerical variables of sociodemographic and clinical characteristics will be made with an independent two-sample t-test for normally distributed variables, and Mann-Whitney U test for non-normally distributed variables. Repeated measure covariance analysis will be applied to reveal the difference between the milk amounts of the mothers between the groups. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

- Between the ages of 18-35,

* Birth after 37 weeks of gestation,
* Caesarean section with regional anesthesia,
* Primiparous,
* No contraindications for breastfeeding (infection, contraindicated drug use, breast problems, etc.),
* Having no health problems (tuberculosis, HIV, cancer, etc.),
* Not using drugs to increase breast milk, vitamins and additional supplements,
* Does not have any problems preventing communication,
* At least primary school graduate,
* Able to speak and understand Turkish,
* Volunteer mothers who agree to participate in the study will be included.

Exclusion Criteria:

* • The baby has contraindications for breastfeeding (galactosemia, congenital anomalies, etc.),

  * Having postpartum complications (bleeding, embolism, etc.),
  * Separated from her baby for any reason after birth (in cases where the mother or baby is referred, hospitalized in intensive care or isolated),
  * Having complications during pregnancy (gestational diabetes, preeclampsia, Rh incompatibility, heart disease, etc.),
  * Tissue integrity deteriorated in the area to be treated,
  * Having lost her baby,
  * Smoking or using alcohol,
  * Those who test positive for Covid-19 will be excluded from the study.
  * Those who want to leave the research at any stage of the research will be excluded from the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
amount of breast milk | The baby will be weighed 8-12 hours after the cesarean section.
  The baby will be weighed before and after breastfeeding. The amount of milk will be calculated according to the difference in weight.
amount of breast milk | Reported the use of baby weighing in postoperative period on 1.days at 8.00-12:00 am.
  The baby will be weighed before and after breastfeeding. The amount of milk will be calculated according to the difference in weight.
amount of breast milk | Reported the use of baby weighing in postoperative period on 1.days at 16.00-20:00 pm.
  The baby will be weighed before and after breastfeeding. The amount of milk will be calculated according to the difference in weight.
amount of breast milk | Reported the use of baby weighing in postoperative period on 2.days at 08.00-16:00 am.
  The baby will be weighed before and after breastfeeding. The amount of milk will be calculated according to the difference in weight.
Visual Analogue Scale by which Mothers Evaluate Lactation Onset Signs | The Visual Analogue Scale, in which the Mothers Evaluate Lactation Onset Symptoms, will be filled in by the mothers between 8-12 hours of the cesarean section.
  Tension, temperature increase and pain in the breasts, which are the signs of starting lactation, will be scored between 0-10. 0 "None", 1-2 "Too little", 3-4 "A little too much", 5-6 "Too much", 7-8 "Too much" and 9-10 "Too much, unbearable" and what is the total score? it will be understood that the higher the lactation onset symptoms, the more
Visual Analogue Scale by which Mothers Evaluate Lactation Onset Signs | The Visual Analogue Scale, in which the Mothers Evaluate Lactation Onset Symptoms, will be filled in by the mothers between in postoperative period on 1.days at 16.00-20:00 pm.
  Tension, temperature increase and pain in the breasts, which are the signs of starting lactation, will be scored between 0-10. 0 "None", 1-2 "Too little", 3-4 "A little too much", 5-6 "Too much", 7-8 "Too much" and 9-10 "Too much, unbearable" and what is the total score? it will be understood that the higher the lactation onset symptoms, the more
Visual Analogue Scale by which Mothers Evaluate Lactation Onset Signs | The Visual Analogue Scale, in which the Mothers Evaluate Lactation Onset Symptoms, will be filled in by the mothers between in postoperative period on 2.days at 08.00-16:00 am
  Tension, temperature increase and pain in the breasts, which are the signs of starting lactation, will be scored between 0-10. 0 "None", 1-2 "Too little", 3-4 "A little too much", 5-6 "Too much", 7-8 "Too much" and 9-10 "Too much, unbearable" and what is the total score? it will be understood that the higher the lactation onset symptoms, the more

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Taşpınar, Prof. Dr., Study Director — aytaspinar@yahoo.com
Locations (1):
- Aydın Adnan Menderes University, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No